CLINICAL TRIAL: NCT03673774
Title: Prognostic Value of Cardiac Output Measured by Impedancemetry in Patients Monitored for Pulmonary Hypertension
Brief Title: Impedancemetry in Patients Monitored for Pulmonary Hypertension
Acronym: HPepic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: RECRUITMENT ISSUES
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/15/7849
Record Dates: First submitted 2018-08-13; First posted 2018-09-17 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; impedancemetry; cardiac output
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardiac impedancemetry (Experimental): Monocentric cohort study, prospective, evaluating the variability of cardiac output measurement by resting and stress impedancemetry as a prognostic factor for PH. Patients are included via the competence center of the PHP of the Midi Pyrenees region. The cardiac output is measured by impedance measurement at rest and during the walking test. The NO / CO coupled transfer measurement is performed at rest. The physician performing the consultation will not know the results of the IPC and these results will not influence the subsequent management.
  The patient will be followed for 18 months as part of the research.
  Interventions: Device: cardiac impedancemetry

INTERVENTIONS:
Device: cardiac impedancemetry — The cardiac output is measured by impedance measurement at rest and during the walking test.

SUMMARY:
Monocentric cohort study, prospective, evaluating the variability of cardiac output measurement by resting and stress impedancemetry as a prognostic factor for Pulmonary Hypertension

DETAILED DESCRIPTION:
Cardiac impedancemetry is a technique that allows an electrical representation of cardiac flows. To do this, 6 electrodes are applied to the thorax and a low intensity and high frequency electrical current is transmitted. The impedance is recorded and the variations of the impedance represent the changes in intra-thoracic volume and thus the volume of systolic ejection. This measurement can be done at rest but also during exercise during the walking test. A test of the NO / CO coupled transfer measurement is also performed.

The devices that will be used in this project are the Physio-Flow® system and Masterscreen NO / CO coupled transfer measurement device

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years and under 80 years
* Patients who have been diagnosed with PAH (group 1 PH according to the Nice 2013 classification) or post-embolic pulmonary hypertension (group 4 PH) under medical treatment;
* HTP incident or prevalent less than 6 months
* Patient coming for follow-up or emergency consultation or hospitalization with a clinical examination and a walking test
* Patient affiliated to a health insurance scheme
* Patient having signed informed consent

Exclusion Criteria:

* Subjects under juridical protections or tutelage measure
* pregnant or lactating woman
* pulmonary hypertension du to cardiac pathology, chronic respiratory disease, or uncertain determinism.
* pulmonary hypertension of group 4 treated surgically or endoscopically.
* pulmonary hypertension incident or prevail for 6 months or more
* contraindication to impedancemetry
* inability to perform a walking test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Measure of cardiac flow variation at 0 month by impedancemetry | 0 month
  The variation of cardiac flow is measured by impedancemetry at rest
Measure of cardiac flow variation at 6 month by impedancemetry | 6 month
  The variation of cardiac flow is measured by impedancemetry at rest

SECONDARY OUTCOMES:
Measure of cardiac flow variation during walking test | 0 month
  The variation of cardiac flow is measured by impedancemetry during walking test
Measure of cardiac flow variation during walking test at 6 month | 6 month
  The variation of cardiac flow is measured by impedancemetry during walking test
Correlation between measurement of capillary blood volume and measurement of cardiac flow | 0 month
  Evaluate the correlation between measurement of capillary blood volume and measurement of cardiac flow by impedancemetry
Correlation between measurement of capillary blood volume and measurement of cardiac flow | 6 month
  Evaluate the correlation between measurement of capillary blood volume and measurement of cardiac flow by impedancemetry
Occurrence of an undesirable event | 18 month
  Collection of undesirable event like : - Deaths (all causes combined), Hospitalization for aggravation of PAH, Progression of the disease or decrease, Unsatisfactory long-term clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Elise Noel-Savina, MD, Principal Investigator — CHU of Toulouse
Locations (1):
- CHU TOULOUSE hospital larrey, Toulouse, Midi-Pyrennée, France